CLINICAL TRIAL: NCT01592214
Title: A Two-Part Phase I Study to Establish and Compare the Safety and Local Tolerability of Two Nasal Formulations of XF-73 for Decolonization of Staphylococcus Aureus: A Previously Investigated 0.5 mg/g Viscosified Gel Formulation Versus a Modified Formulation
Brief Title: Study of the Safety and Local Tolerability of Intranasal Gel Formulations of XF-73
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11-0007; HHSN272201500007I; XF-73
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-07

CONDITIONS: Staphylococcal Infection
Keywords: Staphylococcus aureus, nasal decolonization, XF-73, gel formulation
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Part 1 #2-XF-73 in 2% Klucel® gel, concentration 2.0 mg/g (Experimental): 4 subjects: 2.0 mg/g concentrations of a modified 2% Klucel® gel formulation of XF-73 intranasally to both nares twice in a single day in a volume of 0.3 mL/naris/dose and total daily dose of 2.4 mg.
  Interventions: Drug: XF-73 in 2% Klucel gel
- Part 2 #4-Placebo in 4% Klucel® gel, concentration 0 mg/g (Placebo Comparator): 12 subjects: a placebo in 4% Klucel® gel intranasally to both nares in a volume of 0.3 mL/naris/dose,3 doses 8 hours apart on Day 1 and 2 doses, 12 hours apart on Days 2 to 5. Total daily volume of 1.8 ml on Day 1 and 1.2 ml on Days 2 to 5.
  Interventions: Other: Placebo
- Part 2 # 3-XF-73 in 4% Klucel® gel, concentration 0.5 mg/g: (Active Comparator): 12 subjects: a modified 4% Klucel® gel formulation of XF-73 intranasally to both nares in a concentration of 0.5 mg/g and volume of 0.3 mL/naris/dose in, 3 doses 8 hours apart on Day 1 and 2 doses, 12 hours apart on Days 2 to 5. Total daily volume of 1.8 ml on Day 1 and 1.2 ml on Days 2 to 5; and total daily dose of 0.9 mg on Day 1 and 0.6 mg on Days 2 to 5.
  Interventions: Drug: XF-73 in 4% Klucel gel
- Part 2 #2- XF-73 in 2% Klucel® gel, concentration 2.0 mg/g (Experimental): 12 subjects; a modified 2% Klucel® gel formulation of XF-73 intranasally to both nares in a concentration of 2.0 mg/g and volume of 0.3 mL/naris/dose,3 doses 8 hours apart on Day 1 and 2 doses, 12 hours apart on Days 2 to 5. Total daily volume of 1.8 ml on Day 1 and 1.2 ml on Days 2 to 5; and total daily dose of 3.6 mg on Day 1 and 2.4 mg on Days 2 to 5.
  Interventions: Drug: XF-73 in 2% Klucel gel
- Part 2 #1- XF-73 in 2 % Klucel® gel, concentration 0.5 mg/g (Experimental): 12 subjects: a modified 2% Klucel® gel formulation of XF-73 intranasally to both nares in a concentration of 0.5 mg/g and volume of 0.3 mL/naris/dose, 3 doses 8 hours apart on Day 1 and 2 doses, 12 hours apart on Days 2 to 5. Total daily volume of 1.8 ml on Day 1 and 1.2 ml on Days 2 to 5; and total daily dose of 0.9 mg on Day 1 and 0.6 mg on Days 2 to 5.
  Interventions: Drug: XF-73 in 2% Klucel gel
- Part 1 #1-XF-73 in 2% Klucel® gel, concentration 0.5 mg/g: (Experimental): 4 subjects: 0.5 mg/g concentration of a modified 2% Klucel® gel formulation of XF-73 intranasally to both nares twice in a single day in a volume of 0.3 mL/naris/dose and total daily dose of 0.6 mg.
  Interventions: Drug: XF-73 in 2% Klucel gel

INTERVENTIONS:
Other: Placebo — Placebo: 4% Klucel® gel formulation, concentration 0, total daily volume 1.8 ml, 3 doses 8 hours apart on Day 1 and 1.2 ml, 2 doses 12 hrs apart on Days 2 to 5.
  Arms: Part 2 #4-Placebo in 4% Klucel® gel, concentration 0 mg/g
Drug: XF-73 in 2% Klucel gel — XF-73 in a modified 2% Klucel® gel formulation: Part 1, #1: concentration 0.5 mg/g, twice a day in volume 0.3 mL/naris/dose, total dose 0.6 mg; Part 1, #2: 2.0 mg/g concentration, twice a day in volume 0.3 mL/naris/dose, total dose 2.4 mg; Part 2, #1: Concentration 0.5 mg/g, 3 doses 8 hours apart on Day 1, total volume 1.8 ml, total dose 0.9 mg, 2 doses 12 hours apart on Days 2-5, total volume 1.2 ml and total dose 0.6 mg ; Part 2, #2: 2.0 mg/g, 3 doses 8 hours apart on Day 1, total volume 1.8 ml, total dose 3.6 mg, 2 doses 12 hours apart on Days 2-5,total volume 1.2 ml and total dose 2.4 mg.
  Arms: Part 1 #1-XF-73 in 2% Klucel® gel, concentration 0.5 mg/g:; Part 1 #2-XF-73 in 2% Klucel® gel, concentration 2.0 mg/g; Part 2 #1- XF-73 in 2 % Klucel® gel, concentration 0.5 mg/g; Part 2 #2- XF-73 in 2% Klucel® gel, concentration 2.0 mg/g
Drug: XF-73 in 4% Klucel gel — XF-73 in a 4% Klucel® gel formulation: Part 2 #3: concentration of 0.5 mg/g and volume of 0.3 mL/naris/dose in 3 doses 8 hours apart on Day 1 and 2 doses, 12 hours apart on Days 2 to 5. Total daily volume of 1.8 ml on Day 1 and 1.2 ml on Days 2 to 5; and total daily dose of 0.9 mg on Day 1 and 0.6 mg on Days 2 to 5.
  Arms: Part 2 # 3-XF-73 in 4% Klucel® gel, concentration 0.5 mg/g:

SUMMARY:
This is a Phase I, multi-center, clinical study of XF-73 to evaluate the local (nasal) safety and tolerability of a modified, thinner lower viscosity formulation of intranasal XF-73 in healthy male and female subjects. In addition, the potential for systemic absorption of XF-73 in the modified, thinner lower viscosity and the previously investigated thicker, higher viscosity formulations and their decolonization efficacy in comparison to placebo will be evaluated. Both parts of the study will be double-blinded and Part 2 will also be placebo-controlled. Primary objective is to establish the safety and tolerability of two concentrations of a modified thinner, lower viscosity nasal formulation of XF-73 and to compare them to a previously investigated, thicker, higher viscosity formulation

DETAILED DESCRIPTION:
This is a Phase I, multi-center, clinical study of XF-73 to evaluate the local (nasal) safety and tolerability of a modified, thinner, lower viscosity formulation of intranasal XF-73 in healthy male and female subjects. In addition, the potential for systemic absorption of XF-73 in the modified, thinner, lower viscosity and the previously investigated thicker, higher viscosity formulations and their decolonization efficacy in comparison to placebo will be evaluated. Both parts of the study will be double-blinded, and Part 2 will also be placebo-controlled. Study subjects will be healthy volunteers, male or female, aged 18 - 45 years. The study will be conducted in two distinct parts. In Part 1 of the study 8 healthy male and female subjects, aged 18 to 45 years, will be in two groups of four per formulation will have a study duration of up to 36 days. All subjects will receive intranasal applications of 5,15-bis-[4-(3-Trimethylammonio-propyloxy)-phenyl]-porphyrin dichloride (XF-73). In Part 2 only, subjects will also need to be confirmed as persistent nasal SA carriers (n = 48). (Persistent SA carriage is defined by 3 separate, SA positive cultures from nasal swabs: the first taken at Pre-Screening no more than 12 weeks (84 days). Administration will last five days, being three times a day on Day 1, then twice a day thereafter. Primary objective is to establish the safety and tolerability of two concentrations of a modified thinner, lower viscosity nasal formulation of XF-73 and to compare them to a previously investigated, thicker, higher viscosity formulation. Secondary objectives are to establish whether there is any potential systemic exposure following administration of the two nasal formulations of XF-73 and to evaluate the anti-staphylococcal efficacy of two concentrations of a lower and one of a thicker, higher viscosity nasal formulation of XF-73.

ELIGIBILITY:
Inclusion Criteria:

1. Normal, healthy male or female subjects aged between 18 and 45 years inclusive.
2. For Part 2 only: Normal healthy subjects confirmed to be persistent SA carriers (NOTE: Persistent SA carriage is defined by 3 separate, SA (Staphylococcus aureus) positive cultures from nasal swabs: the first taken at Pre-Screening no more than 12 weeks (84 days) prior to first dosing, a confirmatory swab taken at Screening at least 7 days after Pre-Screening and a final confirmation swab taken on Admission, a day before dosing and at least 7 days after screening. Subjects may be dosed with only two positive swabs while awaiting the result of the third swab obtained on Admission, but dosing will be discontinued in subjects whose Admission swab is found to be negative for SA.
3. Subject must be healthy, in the opinion of the Investigator, as determined by medical history (MH), physical examination (PE), normal nasal examination, and vital signs (VS).
4. Subject's 12-lead electrocardiogram (ECG) must be normal or abnormal not clinically significant as reported by the overreading cardiologist.
5. Subject's clinical laboratory results at Screening must be within the reference range or expanded range.Subjects may undergo a repeat screening test of out-of-range analytes at the discretion of the investigator to confirm a plausible alternative explanation that will be indicated in the source documentation.
6. Any subject having laboratory values outside of the reference range or expanded range at Day -1 but were within the reference or expended range at screening may be enrolled on study. Abnormal urine dipstick values for blood/hemoglobin, nitrite, and leukocyte esterase will not be exclusionary if a microscopic examination of the urine on the same sample or the most recent sample obtained prior to dosing is within the reference or expanded range. Laboratory values outside the reference or expanded range will be assigned to toxicity grade.
7. Subjects who are able and willing to provide written informed consent to participate in the study.
8. Subject agrees to comply with all study requirements.
9. All female subjects of childbearing potential must have a negative serum and urine pregnancy test at Screening and Admission respectively.
10. Subjects who have a body mass index (BMI) >/= 18.5 kg/m^2 and </= 35 kg/m^2.
11. Subject agrees not to participate in another clinical trial at any time during the study period.

Exclusion Criteria:

1. Female subjects who are pregnant or who are lactating.
2. Heterosexually active females of child-bearing potential, defined as being physiologically capable of becoming pregnant, unless they agree to use two of the following acceptable methods of contraception throughout their participation in the study and for at least 12 weeks after the final dose: (a) established use of oral, injected or implanted hormonal contraception, (b) intrauterine Device (IUD or Coil), (c) a female barrier method (diaphragm or cervical/vault cap) and/or (d) condom plus spermicidal cream/gel. Women who are not sexually active (abstinent) but become active must use two of the listed contraceptive methods.
3. Heterosexually active males unless they agree to use two concomitant acceptable methods of contraception throughout their participation in the study and for at least 12 weeks after receiving their final dose of study medication (examples include: vasectomy combined with latex condom with spermicide, latex condom with spermicide combined with a female partner who practices an acceptable method of contraception as indicated above); Men who are not sexually active (abstinent) but become active must use two of the listed contraceptive methods. Subjects who currently have or have had any acute illness within the past two weeks.
4. Subjects who currently have or have had within the past two weeks a poorly controlled chronic illness(anemia, thrombocytopenia, or coagulation disorders), cancer, infection, or any other clinically significant disorder.
5. Subjects who currently have or have had an autoimmune disease.
6. Subjects who have had within the past two weeks a symptomatic upper respiratory tract infection, nasopharyngitis, influenza or condition involving increase in nasal secretion such as seasonal or chronic, allergic rhinitis. Additionally, any subject with history of atopy/allergies within the past 30 days will be excluded.
7. Subjects who have had been diagnosed with a concussion within the past two years.
8. Subjects with a history of serious psychiatric condition (depression, bipolar disorder, schizophrenia, suicidal ideation, or suicide attempts) or receiving two concomitant medications for the treatment of a psychiatric disorder or hospitalized for the treatment of a serious psychiatric disorder within six months of participation in the study.
9. Subjects with known skin photosensitivity.
10. Subjects with a personal or family history of porphyria.
11. Subjects with any open wound, lesion, inflammation, erythema, or infection affecting the nostrils, nose, upper lip, and area of skin close to the nose, including herpes simplex lesions and discoid lupus.
12. Subjects with a history of abnormal bleeding, bruising, frequent nosebleeds, or the diagnosis of von Willebrand disease.
13. Subjects with nasal polyps or significant anatomical nasal abnormality. Patients with deviated septa will be allowed in the study, provided the principal investigator does not deem a deviation to be of significant medical consequence. An ENT(Ear, Nose and Throat) specialist will be available for consult as needed.
14. Subjects with a history of nasal surgery, including cauterization, in the last 6 months.
15. Subjects with a history of multiple episodes [>3] of epistaxis within the 12 months prior to screening.
16. Subjects with in situ nasal jewelry or open nasal piercings.
17. Subjects with a known clinically significant history of atopy or hypersensitivity to any drug or latex or to ingredients of the nasal gel (such as benzalkonium chloride or other quaternary ammonium disinfectants) or to drugs related to XF-73.
18. Subjects known to have dermal sensitivity to chlorhexidine gluconate (CHG).
19. Subjects who have smoked within the month prior to screening.
20. Subjects who have been treated with or have taken any prescribed or over-the-counter medication daily for the last 14 days, with the exception of hormonal contraceptives or hormone replacement therapy.
21. Subjects who have taken or used topical or systemic antibiotics within the month prior to screening.
22. Subjects who have received an immunization within 30 days prior to screening.
23. Subjects with a history of drug or alcohol abuse in the last 12 months or who have a positive urine drug test for substances of abuse (amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine metabolites, opiates, phencyclidine [PCP]) or alcohol.
24. Subjects who are known to have serum hepatitis, or who are carriers of the hepatitis B surface antigen(HBsAg) or hepatitis C (HCV) antibody, or who have a positive result to the test for human immunodeficiency virus (HIV) antibodies.
25. Subjects who have participated in a drug or vaccine clinical trial within the last month.
26. Subjects who have been exposed to XF-73 as part of a previous clinical trial.
27. Presence of any other condition or laboratory result that, in the opinion of the investigator would jeopardize the safety or rights of a subject participating in the trial or would render the subject unable to comply with the protocol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The local (nasal and nasal passage) and systemic safety and tolerability of XF-73 following nasal administration in healthy male and female subjects | Day 1 through Day 8 (Part 1) and Day 1 through Day 14 (Part 2)

SECONDARY OUTCOMES:
In the Part 2 of the study, anti-staphylococcal activity will be investigated, activity will be assessed as the presence or absence of SA and by quantification of the level of colonization | Part 2: Enrollment, Day 1 through Day 6 and Day 14.
The efficacy of the modified formulation of XF-73 and of the previous formulation on nasal load of S. aureus after daily treatment with XF-73 for five days as compared to placebo (in Part 2 of the study only). | Part 2: Enrollment, Day 1 through Day 6 and Day 14.
The pharmacokinetics (PK) of XF-73 following nasal administration of two concentrations of a modified formulation (in both parts of the study) and a single concentration of a previously investigated formulation (in Part 2 of the study). | Part 1: 0 hr, at 15, 30 min, 1, 2, 4, 8, 12 hr after each dose. Part 2 within 15 min before 1st dose, 30, 240, 480 min after 1st dose. Day 3: 30 min after 1st dose; Day 5: within 15 min before 1st dose, 30, 240 min after.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Anaheim Clinical Trials - Phase I Clinical Pharmacology Unit, Anaheim, California
  - Case Western Reserve University - Case Medical Center - Infectious Disease & HIV Medicine, Cleveland, Ohio